# **COVER PAGE**

STUDY TITLE: Study of the Families Moving Forward Website Behavioral Intervention for Teachers of Students With Fetal Alcohol Spectrum Disorder

NCT05986565

**DOCUMENT DATE: 10/24/2023** 

## Pilot Trial of the FMF Connect Teacher Companion Website Principal Investigators – Christie Petrenko and Cristiano Tapparello

### 1. PURPOSE OF STUDY

The purpose of this study is to evaluate feasibility of the FMF Connect Teacher Companion website and study design through a pilot trial. Specifically, we will investigate 1) intervention feasibility and 2) study design acceptability. Intervention feasibility includes technological feasibility of the website, acceptability of the website, and typical usage patterns. Study design acceptability includes enrollment and attrition rates, acceptability of randomization and control condition, assessment acceptability and sensitivity, optimal intervention length, and predictors of attrition

## Our hypotheses are:

- 1) the website will be technologically functional and acceptable to users, and users will show a moderate level of engagement with the website as evidenced by at least one hour per week of use.
- 2) the study design and assessments will be acceptable, the study will have sufficient enrollment to meet recruitment targets, and attrition will be predicted by teacher type (general education teacher) and teacher level of experience with FASD (teachers with less experience will be more likely to remain in the study).

This study is a pilot trial. Pilot trials are indicated when there is little information using a specific intervention technique in a certain population or the target population has been shown to need unique consideration of the topic (Bowen et al., 2009).

### 2. BACKGROUND AND RATIONALE

Fetal alcohol spectrum disorders (FASD) affect an estimated 1.1-5% of children in the US (May et al., 2018) and can impact various aspects of neurodevelopment, including executive functioning, behavior, and academic performance. Although the majority of individuals with FASD are not intellectually disabled (Mattson et al., 2011), children with FASD perform lower than nonexposed individuals in academics (Crocker et al., 2015; Glass, 2016; Howell et al., 2006; Jirikowic et al., 2008). Without appropriate support, deficits in executive functioning and self-regulation may lead to difficulty organizing materials, planning, and sustaining attention as well as emotional and behavioral dysregulation. Teachers often lack understanding of FASD, leading to ineffective strategies and frustration. Lack of awareness and insufficient training on FASD in the school system creates significant barriers to services for children with FASD (Dybdahl & Ryan, 2009; Koren et al., 2010; Millar et al., 2017; Ryan & Ferguson, 2006; Ryan et al., 2006). Parents often report struggling to obtain services and supports for their children in schools and describe having to educate teachers and staff about FASD (Petrenko et al., 2014; Petrenko et al., 2020; Ryan & Ferguson, 2006; Ryan et al., 2006).

In-person trainings are limited in reach, while a digital intervention delivered via the internet can provide broader access and flexibility. The Families Moving Forward (FMF) Program is a scientifically-validated behavioral consultation program developed at Seattle Children's Research Institute/University of Washington by Heather Carmichael Olson and colleagues (Bertrand, 2009; Olson & Montague, 2011; Petrenko et al., 2017). It is usually delivered in person or via telehealth by trained specialists. It is designed for caregivers of

children with FASD and includes an in-person, targeted school consultation in which a specialist works with school staff to educate them on FASD, build a more positive home-school relationship, and discuss ways to better support the student. Educating teachers to increase their knowledge and awareness of FASD is hypothesized to help them to modify their attributions of the student's behavior and use more effective behavioral strategies, leading to improved self-efficacy and student-teacher relationship.

Given lack of widespread awareness of FASD, stigma. and numerous systems barriers (Petrenko et al., 2014; Roozen et al., 2020), many families in need of evidence-based intervention do not receive it. To address this need, the FMF Connect mobile Health (mHealth) app was derived from the standard FMF Program to directly provide caregivers with easily accessible, self-directed, evidence-based content and resources. In development and initial feasibility trials of FMF Connect, parents stressed the importance of materials or interventions for teachers (Petrenko et al., 2020; 2021). The FMF Connect Teacher Companion website was developed using the ADAPT-ITT framework (Wingood & Clemente, 2008) to address this need. It includes materials and exercises from the FMF Program and FMF Connect which have been adapted to teachers, incorporating a teacher needs assessment and a Teacher Advisory Board.

The current study will pilot the FMF Connect Teacher Companion website to determine technological acceptability and feasibility of study design and methods to inform a future RCT. This trial is designed using best practices in pilot/feasibility trials (Lancaster et al., 2004; Eldridge et al., 2016) and will follow the CONSORT extension for pilot trials in reporting and publishing (Eldridge et al., 2016). Aligning with the FMF model, the Teacher Companion website is the next logical step to disseminate this empirically-validated treatment and will complement FMF Connect in building a scalable and accessible network of support for children with FASD and their families.

The FMF Connect Teacher Companion website will increase accessibility of evidence-based materials on FASD for teachers, which is particularly critical for rural and other underserved populations. Websites can be easily accessed across a number of platforms including a mobile phone, tablet, laptop, or desktop computer, necessary for teachers who may work in a variety of settings, and are less likely to use a mobile phone in the classroom. This increased accessibility will allow teachers to more successfully manage behavior and support learning of students with FASD and will decrease barriers to quality care and services faced by many caregivers of children with FASD (Petrenko et al., 2014; Roozen et al., 2020; Ryan et al., 2006). This project will advance scientific knowledge relating to teacher awareness, perceptions, behavioral strategies, and self-efficacy related to FASD. It will also address a need for a systematically developed intervention which can be tested and improved through rigorous and reproducible research. Although some teacher resource websites for FASD exist, this will be the first empirically-derived and tested digital teacher intervention specific to FASD.

### 3. ADMINISTRATIVE ORGANIZATION

This study is led by Drs. Christie Petrenko and Cristiano Tapparello. Dr. Petrenko is faculty at Mt. Hope Family Center and has appointments in the departments of Psychology and Pediatrics. Dr. Tapparello is faculty in the department of Electrical and Computer Engineering. They will oversee all research staff, implementation of human subjects' protections, and data collection, management, analysis, and reporting.

All data collection will be through our research team at the University of Rochester. Participants

will be recruited online and complete informed consent, screening, and survey through our REDCap database, hosted at the University of Rochester. Interview data will be collected via HIPAA-complaint Zoom. Additional data will be collected through the FMF Connect Teacher Companion website, developed and managed by our team and hosted on a URMC-managed Azure account.

#### 4. STUDY DESIGN

The study design is a 2-parallel arm, staggered design pilot RCT. All subjects will complete baseline assessments. Then they will be randomly assigned to either Group 1) Website, or Group 2) Delayed treatment control. Group 1 will receive access to the website immediately. After six weeks, both groups will complete Timepoint 2 assessments. Selected participants will complete a qualitative interview about their experience using the website. After completion of Timepoint 2 assessments, Group 2 will receive access to the website (Group 1 will retain access to the website). After an additional six weeks, both groups will complete Timepoint 3 assessments and the study will conclude.

Assessments will include measures of FASD knowledge, teacher self-efficacy, teacher attributions and behavioral strategies, and satisfaction with the technology and study. Website usage data will be collected using Azure Application Insights (feature that can be enabled on our URMC-managed Azure account). Participants will be assigned to groups using simple randomization using manual 50/50 chance randomization.

#### 5. SUBJECT POPULATION

The study population will be U.S. teachers of grades K-5. We will aim to enroll 90 participants to achieve a final sample size of 50, assuming a 45% attrition rate (consistent with recent 3-timepoint online studies in our lab). Additional participants will be enrolled if attrition is greater than anticipated.

#### 6. INCLUSION AND EXCLUSION CRITERIA

Inclusion Criteria

Subjects must:

- Be an educational professional currently actively employed in a school setting in the United States
- Be above the age of 18 years old
- Have direct, consistent contact with a student with a diagnosed fetal alcohol spectrum disorder (FASD) or confirmed prenatal alcohol exposure (PAE) between the ages of 5-12, (i.e. grades K to 5) in a special or general education classroom
- Have reliable access to the Internet
- Be able to consent for themselves

Exclusion criteria:

Subjects will be excluded if:

- They are unable to read English
- They do not have direct, consistent contact with a student with a diagnosed FASD between ages 5-12 (e.g., substitute teacher, principal)

#### 7. RECRUITMENT METHODS

Subjects will be recruited nationally through a number of sources:

- In order to directly target teachers in under-resourced areas, we will identify low-income school districts using the Teacher Cancellation Low Income (TCLI) directory. This directory includes schools identified as low-income for the purposes of federal aid. We will randomly select districts in different states from this directory and reach out to administrative personnel about the study. If interested and willing, they will send out information about the study to the teachers in the district.
- We will also recruit via parent participants involved in trials of the FMF Connect app, all of whom have children with confirmed PAE or FASD. Parents with a child between the ages of 5-12 who have consented to receiving information about future research will receive an email informing them about the Teacher Companion website trial. This email will encourage them to share recruitment materials with their child's teacher for the upcoming year if interested. Teachers can then contact the study team if they would like to participate and will be encouraged to forward to any other eligible teachers.
- If these two methods do not prove adequate in recruiting sufficient and diverse subjects, we will target teachers and school staff through national email newsletters and social media forums specific to teachers. We will also send recruitment materials to disability- and FASD-specific networks such as the University Centers for Excellence in Developmental Disabilities (UCEDD) email listserv and FASD special interest groups. Finally, we will engage colleagues in the FASD field to send recruitment materials to their networks to recruit teachers who have a student with FASD.

### 8. CONSENT PROCESS

Given this research is no greater than minimal risk and involves procedures for which written consent is normally not required outside of the research context (e.g., survey responses, website usage), we are requesting a waiver of documentation of consent. There is also not an easy way to verify participant identify for written eConsent without creating an additional step for participants involving communication with research staff through another method (e.g., email, phone).

Subjects who are interested in participating in the study will be directed to the REDCap Screening Module where they will view the Study Information Sheet. After reviewing the Study Information sheet, they will be asked several questions assessing their understanding of the information. All subjects will be given the option to download a copy of the Information Sheet for their records.

The study coordinator's contact information will also be presented if participants want to contact the coordinator with questions while reading the document. The study coordinator will document contact in the study contact log in REDCap. Additional items will screen for eligibility and obtain contact information.

The primary identifying information collected as part of this study are participant contact information in the REDCap Screening Module. This contact information would allow us to

contact participants in several anticipated scenarios, such as: if they indicate they have questions about the study, they provide inconsistent information we need to clarify, or to send them surveys or schedule interviews.

Identifying information will be stored separately from other de-identified data sources.

After reviewing the information sheet and completing comprehension questions, participants will be directed in REDCap to answer screening questions to assess eligibility for the study (see Screening Form). If eligibility criteria clearly aren't met (e.g., doesn't have a student with FASD), participants will be informed immediately that they aren't eligible and the module will end. Screening data will be maintained for ineligible participants to aid in clinical trial reporting requirements (e.g., documenting numbers screening, eligible vs. ineligible, and reasons).

This study is funded by the National Institute of Health (NIH). A Certificate of Confidentiality is automatically included as part of the notice of award. Language regarding the Certificate of Confidentiality is included in the consent documents.

Due to an increase in fraudulent participants across studies in our lab, we have developed a labwide guide to prevent, detect, and systematically manage fraudulent participants (see uploaded). For this study, if "red flags" (e.g., common email formula, unusual emails; see lab-wide guide for other examples) are identified by research staff, they will follow lab scripts to withdraw the participant.

### 9. STUDY PROCEDURES

After informed consent, participants will be asked to complete screening questions to assess for eligibility criteria. Subjects who are not eligible will be told immediately and the module will end. Subjects who are eligible will be randomized to either Group 1 (Website) or Group 2 (Delayed Treatment Control). Randomization will be completed using manual 50/50 chance randomization. After randomization, subjects will complete the remaining baseline surveys (see details on the assessment battery below).

Once baseline surveys are complete, subjects in Group 1 will receive immediate access to the website. After 6 weeks, all subjects will be re-contacted to complete timepoint 2 surveys. User implementation data will be gathered through the website. To further assess acceptability, satisfaction, and barriers and facilitators of website use, selected participants will complete qualitative interviews over HIPAA-complaint Zoom or telephone. Interviews will be recorded and later transcribed verbatim. Participants will be selected for interviews based on patterns of website usage, personal demographics such as race, ethnicity, job title, and years of experience, and school geographic setting. A total of 5 participants will be interviewed from Group 1 at Timepoint 2.

After completion of Timepoint 2 assessment, Group 2 will receive access to the website (Group 1 will retain access to the website). After another six weeks, all subjects will complete Timepoint 3 assessments. A total of 5 participants will be interviewed from Group 2 at Timepoint 3, selected using the same procedure as for Timepoint 2.

The study coordinator will email participants to the email they provided to inform them they have access to the website and alert them to their login information.

Participants will be prompted to complete surveys upon reaching each timepoint via automated

invitation sent to the email they provided in REDCap. If they do not complete the surveys within three days, they will be sent another email reminder. If they do not complete the surveys within a week after the first reminder, they will be called by the study coordinator.

The project coordinator will track participants in REDCap once enrolled and will facilitate timely completion of research assessments. All participants will be encouraged to complete assessments, regardless of their level of engagement with the FMF Connect Teacher Companion website. Actual user data from the website (whether minimal or extensive) will be important in addressing study aims.

Study Assessment Battery

| Measure | Number<br>Items | Baseline | T2 | Т3 |
|---|---|---|---|---|
| Screening and Demographics Measure:<br>This includes both the screening<br>questions and demographics including<br>information about teaching experience<br>and setting | 39 | X | | |
| FASD Knowledge survey: This was adapted from FMF Connect trials and assesses knowledge about FASD | 28 | X | X | X |
| Perceived Self-Efficacy: The Teacher<br>Self Efficacy Scale (TSES) measures<br>teachers' sense of self-efficacy in<br>teaching and supporting students in the<br>classroom | 10 | X | X | X |
| Behavioral Attributions: Attributions are measured by the Reasons for Children's Behavior (RCB) across seven subscales of behavior and willful or ability-based attributions. | 30 | | X | X |
| Behavioral Strategies: The Behavioral Strategies measure was co-normed with the RCB and assesses opinions about common behavioral strategies in the classroom | 36 | X | X | X |
| Time spent on student: These questions assess how much time on average the teacher spends planning for their student with FASD. | 3 | X | X | X |
| Study Design Feasibility and<br>Acceptability: The Study Experiences<br>Survey (SES) was developed for this<br>study and assesses participants'<br>experiences with the study procedures | 10 | | X | |
| Program Satisfaction: The Mobile | 32 | | Group 1 | X |

| Application Rating Scale – User<br>Version (uMARS) assesses<br>functionality, usefulness, and<br>helpfulness of technology and<br>information. It is originally used for<br>apps but has been adapted for a<br>website. | | | | |
|---|---|---|---|---|
| Qualitative Interview on User<br>Experience: This is a 30-45 semi-<br>structured interview assessment<br>participants' experiences of using the<br>website and participating in the study<br>(see uploaded questioning route) | N/A | | Group 1 | Group 2 |
| Total number of items at each timepoint | | 116 | 149 (Group 1)<br>117 (Group 2) | 139 |

<u>Qualitative Interview</u>. The semi-structured questioning route will cover the following topics: 1) overall impressions of the FMF Connect Teacher Companion website; 2) experience using the website (both facilitators and barrier of use); and 3) perceived impact on their teaching and classroom experience. Interviews are expected to last about 30-45 minutes.

<u>FMF Connect Teacher Companion website</u>. The FMF Connect Teacher Companion website is designed to offer teachers evidence-based education about FASD and strategies to support students with FASD. It is adapted from the FMF Program and FMF Connect, evidence based interventions to support caregivers of children with FASD. The FMF Program and FMF Connect aim to improve caregivers' efficacy and satisfaction as a parent, efficacy, attributions for their child's behavior, and the parent-child relationship. This study will test if the FMF Connect Teacher Companion website if feasible and acceptable, and measure its preliminary effect on these outcomes in teachers.

Usage data from the website will be collected using Azure Application Insights. Application Insights allows to identify website utilization patterns like, for example, number of active users, number of sessions per user, or specific features that the participants use the most.

#### 10. AUDIO/VIDEO RECORDINGS

Qualitative interviews will be recorded using HIPAA-complaint Zoom. Research staff will be at Mt. Hope Family Center when completing interviews, using UR computers. Recordings will be uploaded from the local machine as soon as possible to a URMC Box folder for this project managed by the IT team at Mt. Hope Family Center. Only research staff involved on this project will have access to recordings. Recordings will then be transcribed verbatim by research staff. After all transcripts have been rechecked, audio and video recordings will be deleted.

### 11. RISKS TO SUBJECTS

Participants may experience psychological risks associated with participation in this study, such as discomfort or boredom in answering questions or providing feedback about the website. There is also a risk of loss of confidentiality. All data collected for the proposed

research study will be kept confidential to the extent allowed by law. Although it is unlikely given the nature of this study, if participants disclose that someone is being maltreated or is a danger to self or others, research staff will need to break confidentiality to make a report to the appropriate authority to ensure safety, as mandated by law. We believe that all identified risks are reasonable given the proposed procedures for protecting against risk.

## **Protections Against Risks**

To minimize risk associated with psychological discomfort, participants will be given the option to skip questions they feel uncomfortable answering. Multiple procedures will be implemented to protect participant confidentiality. In terms of data storage and management, any hard copy data will be secured in locked file cabinets within locked offices, available only to program staff. Electronic data will be stored on URMC managed Box folder for this project, and only project staff with appropriate permissions will be able to access the data. Forms with identifying information will be separated from the data collected and only subject numbers will be retained in data analysis files.

Multiple levels of protection will be put in place to reduce the risk of loss of confidentiality for data collected through the website. Collected data will be stored using a random code that will not allow direct identification of a particular subject, while any data that identify the user will be stored separately. All the connections with the website, as well as connections between the website and the database, will use state of the art authentication and encryption algorithms (e.g., HTTS, SSL and TLS). The Cloud architecture and services will be built and are managed by Dr. Tapparello, under a University-managed Azure account, and in compliance with University policy. Security and Benchmark compliance reports will be received and reviewed by Dr. Tapparello. Access to the data stored on the Cloud will be restricted, access to the data with be logged and backups will be created to allow the users to restore them if/when necessary. Appropriate policies will be set up so that users will be able to add and modify their own data but will be prevented from viewing and modifying other users' data. Unique login credentials will be provided to each participant and will be required to access the content of FMF Connect Teachers companion website. No personal data will be stored by the website on the participant's device.

All information obtained for research will be kept strictly confidential (as allowed by law) by research staff. Participants will be told about all exceptions (e.g., child/dependent adult abuse, harm to self or others) to confidentiality during the consent process. Project staff will be closely supervised by Dr. Petrenko and instructed on confidentiality, including what information is confidential, the limits of confidentiality, and to whom to report concerns.

The FMF Connect Teacher Companion website is viewed as a "value-added" intervention. Participants can continue to seek information on FASD elsewhere or use their preferred behavior management strategies. The alternative to participating in this study is not to participate.

## 12. POTENTIAL BENEFITS TO SUBJECTS

Participants may not experience any direct benefits from participating in this study. However, participants in prior FASD research studies at MHFC have commented on how they value and derive personal satisfaction in participating in research to increase knowledge

about this under-recognized condition and effective strategies to benefit other people with FASD. It is also possible, although not guaranteed, that subjects might derive benefit from using the FMF Connect Teacher Companion website. Possible benefits may include improved self-efficacy, increased knowledge about FASD, and improved classroom management and teaching.

## 13. COSTS FOR PARTICIPATION

There are no costs to participate.

## 14. PAYMENT FOR PARTICIPATION

Subjects will receive \$25 upon completion of assessments at each timepoint. Those who are selected for and complete an interview will receive an additional \$25. Payments will be gift cards. If a participant withdraws from the study they will receive payment for the timepoints they did complete but not for any future timepoints.

### 15. SUBJECT WITHDRAWALS

Subjects will be advised during the consent process that they have the right to withdraw from the study at any time without prejudice. They can choose to use the website as much as they want (or not at all). We are interested in obtaining survey data as well as feedback about the user experience from as many participants as possible, including those who chose not to use the website or found it hard to navigate. This information is useful in identifying ways to improve the website and facilitate user engagement.

Subjects will not be withdrawn without their consent unless they meet the criteria outlined in the Fraudulent Participant Protocol (see uploaded). Subjects who are withdrawn under this protocol will be replaced and will not count toward final enrollment numbers. Subjects can choose not to complete any or all of the study assessments. They can also completely withdraw from the study with no future contact if they choose. In this case, any data they have previously provided may be used in analyses.

### 16. PRIVACY AND CONFIDENTIALITY OF SUBJECTS AND RESEARCH DATA

All data will be used solely for research purposes and will be securely locked in designated file cabinets, URMC managed Box folder dedicated to project, Project REDCap database, and an encrypted, HIPAA-complaint Cloud database (Azure; for data collected via the website; see above). Identifying information will be stored separately from other data, which will be stored by research ID number. Multiple procedures will be implemented to protect participant data collected through the website, which are further detailed in the section "Protections Against Risks" and Data Security Assessment form. Only senior key personnel and project research staff will have access to the data.

The following table summarizes the project data flow. MHFC IT will set up and manage permissions for URMC Project Box folder. Only project staff will have access to REDCap and Box folders.

| Data Element | How Data<br>Collected | Where Data is Stored | How Data is Managed |
|---|---|---|---|
| Information Sheet, | REDCap | REDCap, | MHFC IT; Project Staff |

| Screening Survey, Contact Information | | Back-ups<br>URMC Box | |
|---|---|---|---|
| Baseline (T1) Surveys, Timepoint 2 surveys, Timepoint 3 surveys | REDCap | REDCap,<br>Back-ups<br>URMC Box | MHFC IT; Project Staff |
| Follow-up Interview | Zoom | URMC Box | MHFC IT; Project Staff; Audio/video data is transcribed verbatim; audio/videos deleted once transcript verified |
| FMF Connect<br>Teacher Companion<br>website usage data<br>and User's inserted<br>data | Website<br>and Azure<br>services | URMC-<br>managed<br>account on<br>Azure | Access is restricted to authorized individuals and every access to the data will be logged, data is encrypted in transit and at rest. Azure account is set up in compliance with UR/URMC policies and monitored by ISD. |

### 15. DATA / SAMPLE STORAGE FOR FUTURE USE

All data (de-identified and identifying) will be securely stored locally for an indefinite period. De-identified and identifying information will be stored separately as detailed above. Novel research questions may arise in the future that this important dataset could answer. Retaining identifying information would facilitate contacting individuals (subsequent to new IRB approval) to see if they would be interested in participating in follow-up research. MHFC has well-established data security procedures in place for long-term storage and maintenance of data. Only approved project staff will have access to data.

## 16. DATA AND SAFETY MONITORING PLAN

Because the research involves the provision of a website-based intervention for teachers, the risk for a serious adverse event due to provision of the intervention is low. Adverse events that could occur include adverse events in the classroom involving students with FASD such as aggression or violence towards others, maltreatment, self-harm or suicidality, or threats of violence to others or to the school. However, these occurrences are unlikely to be a direct consequence of participation in the proposed research or intervention.

Dr. Petrenko will assume ultimate responsibility for the safety and well-being of research participants and the integrity of data collected. Dr. Petrenko has conducted several RCTs on interventions for caregivers of children with FASD. She is a licensed psychologist in the state of New York and is involved in other clinical and research activities at MHFC where maltreatment and suicidality are commonly reported.

The well-being of participants will be monitored throughout the course of the proposed research. If there are concerns regarding a participant during interactions with research staff, staff will immediately contact Dr. Petrenko for consultation and a plan will be developed to address the concerns raised. Additionally, because MHFC provides other treatment programs, there are other back-up clinical supervisors available for consultation for

immediate needs. A phone tree will be established, similar to other projects at MHFC, and will be provided to research staff. Dr. Petrenko will meet with research staff at least weekly to provide supervision and will assess participant well-being. Dr. Petrenko will consult with other co-Investigators and clinical staff at MHFC, as appropriate, to address participant well-being concerns.

The IRB will be notified immediately of any adverse events via telephone and submission of a "University of Rochester Serious Adverse Event Report". Such events would also be reported to NICHD. Ethically, we are committed to ensuring the welfare of participants. Any significant mental health or safety issues detected during the conduct of this investigation will be discussed with participants and options for the receipt of services presented.

#### 17. DATA ANALYSIS PLAN

Qualitative Interview Data: Data will be analyzed thematically to understand users' experiences with the FMF Connect Teacher Companion website and research trial. Thematic analysis focuses on identifying patterns or themes within the data. Consistent with the approach advocated by Miles, Huberman, and Saldana (2014), research team members will first familiarize themselves with the data, iteratively reviewing each transcript, and independently assigning initial codes ("first-level coding"). The team will then come together and discuss, operationalize, and refine each code. We will then generate "second-level codes" which consider categories or deeper meanings among first-level codes. During this process we will examine interrelationships and networks among codes and build a preliminary thematic framework. Transcripts will then be recoded and codes refined through further discussion and consensus, as needed. Participant and group "fit" with the framework will also be assessed, with confirmatory and disconfirmatory evidence for the model examined. Participant matrices may also be utilized to examine variance in themes across participants and key demographic factors, pre-post intervention change, or usage patterns. interviews will be coded using qualitative content analysis.

<u>Quantitative Data Analyses</u>: Quantitative analyses will be largely descriptive, as appropriate for pilot trials (Lancaster et al., 2004) and will include effect sizes and 95% confidence intervals of the following measures in the assessment battery:

- FASD Knowledge survey
- Attributions and Behavioral Strategies
- Perceived Self-Efficacy (TSES)
- Study Design Feasibility and Acceptability (SES)
- Program Satisfaction (uMARS)

The below table summarizes how each analysis will address each sub-aim of the current study.

| Aim | Evaluated Using |
|---|---|
| Intervention Feasibility | |
| • technological functionality | uMARS means/standard deviations; website crash reports; user experience interviews |

| • acceptability of website | uMARS means/standard deviations; user |
|---|---|
| | experience interviews |
| • typical usage patterns | Website usage data, including frequency, |
| | length, and timing of use |
| Study Design Acceptability | |
| <ul> <li>enrollment and attrition rates</li> </ul> | N consented; N with complete data; rate of |
| | attrition |
| <ul> <li>acceptability of randomization and control</li> </ul> | SES means/standard deviations; user |
| condition | experience interviews |
| <ul> <li>assessment acceptability and sensitivity</li> </ul> | Rate of assessment completion; pre-post |
| | effect sizes and 95% confidence intervals |
| • optimal intervention length | Website usage patterns |
| <ul> <li>predictors of attrition</li> </ul> | Rate of attrition; demographic and baseline |
| | variables |

#### 18. REFERENCES

- Bertrand, J., & Interventions for Children with Fetal Alcohol Spectrum Disorders Research Consortium. (2009). Interventions for children with fetal alcohol spectrum disorders (FASDs): overview of findings for five innovative research projects. Research in developmental disabilities, 30(5), 986-1006.
- Bowen, D. J., Kreuter, M., Spring, B., Cofta-Woerpel, L., Linnan, L., Weiner, D., ... & Fernandez, M. (2009). How we design feasibility studies. American journal of preventive medicine, 36(5), 452-457.
- Crocker, N., Riley, E. P., & Mattson, S. N. (2015). Visual-spatial abilities relate to mathematics achievement in children with heavy prenatal alcohol exposure. Neuropsychology, 29(1), 108.
- Dybdahl, C. S., & Ryan, S. (2009). Inclusion for students with fetal alcohol syndrome: Classroom teachers talk about practice. Preventing School Failure: Alternative Education for Children and Youth, 53(3), 185-196.
- Eldridge, S. M., Chan, C. L., Campbell, M. J., Bond, C. M., Hopewell, S., Thabane, L., & Lancaster, G. A. (2016). CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ, 355.
- Glass, L. (2016). Characterizing Reading Ability in Children with Prenatal Alcohol Exposure (Doctoral dissertation, UC San Diego).
- Howell, K. K., Lynch, M. E., Platzman, K. A., Smith, G. H., & Coles, C. D. (2006). Prenatal alcohol exposure and ability, academic achievement, and school functioning in adolescence: a longitudinal follow-up. Journal of Pediatric Psychology, 31(1), 116-126.
- Jirikowic, T., Olson, H. C., & Kartin, D. (2008). Sensory processing, school performance, and adaptive behavior of young school-age children with fetal alcohol spectrum disorders. Physical & occupational therapy in pediatrics, 28(2), 117-136.
- Koren, G., Fantus, E., & Nulman, I. (2010). Managing fetal alcohol spectrum disorder in the public school system: A needs assessment pilot. Journal of Population Therapeutics and Clinical Pharmacology, 17(1).
- Lancaster, G. A., Dodd, S., & Williamson, P. R. (2004). Design and analysis of pilot studies:

- recommendations for good practice. Journal of evaluation in clinical practice, 10(2), 307-312.
- Mattson, S. N., Crocker, N., & Nguyen, T. T. (2011). Fetal alcohol spectrum disorders: neuropsychological and behavioral features. Neuropsychology review, 21(2), 81-101.
- Miles, M. B., Huberman, A. M., and Saldana, J. Qualitative data analysis: A methods sourcebook, third edition, Los Angeles, CA: SAGE Publications Inc, 2014.
- Millar, J. A., Thompson, J., Schwab, D., Hanlon.Dearman, A., Goodman, D., Koren, G., & Masotti, P. (2017). Educating students with FASD: linking policy, research and practice. Journal of Research in Special Educational Needs, 17(1), 3-17.
- Olson, H. C., & Montague, R. A. (2011). An innovative look at early intervention for children affected by prenatal alcohol exposure. Prenatal alcohol use and FASD: Assessment and new directions in research and multimodal treatment, 64-107.
- PA Harris, R Taylor, BL Minor, V Elliott, M Fernandez, L O'Neal, L McLeod, G Delacqua, F Delacqua, J Kirby, SN Duda, REDCap Consortium, The REDCap consortium: Building an international community of software partners, J Biomed Inform. 2019 May 9 [doi: 10.1016/j.jbi.2019.103208]
- PA Harris, R Taylor, R Thielke, J Payne, N Gonzalez, JG. Conde, Research electronic data capture (REDCap) A metadata-driven methodology and workflow process for providing translational research informatics support, J Biomed Inform. 2009 Apr;42(2):377-81.
- Petrenko, C. L., Pandolfino, M. E., & Robinson, L. K. (2017). Findings from the families on track intervention pilot trial for children with Fetal Alcohol Spectrum Disorders and their families. Alcoholism: Clinical and Experimental Research, 41(7), 1340-1351.
- Petrenko, C. L., Parr, J., Kautz, C., Tapparello, C., & Olson, H. C. (2020). A Mobile Health Intervention for Fetal Alcohol Spectrum Disorders (Families Moving Forward Connect): Development and Qualitative Evaluation of Design and Functionalities. JMIR mHealth and uHealth, 8(4), e14721. PMCID: PMC7171567
- Petrenko, C. L., Tahir, N., Mahoney, E. C., & Chin, N. P. (2014). Prevention of secondary conditions in fetal alcohol spectrum disorders: identification of systems-level barriers. Maternal and child health journal, 18(6), 1496-1505.
- Petrenko, C.L.M., Kautz-Turnbull, C., Roth, A., Tapparello, C., Demir, U., & Carmichael Olson, H. (Under review). The Families Moving Forward Connect Mobile Health Intervention for Caregivers of Children with Fetal Alcohol Spectrum Disorders: Findings from Beta-Testing Within a Systematic User-Center Design Approach [Manuscript submitted for publication]. Mt. Hope Family Center, University of Rochester.
- Roozen, S., Stutterheim, S. E., Bos, A. E., Kok, G., & Curfs, L. M. (2020). Understanding the social stigma of fetal alcohol spectrum disorders: From theory to interventions. Foundations of Science, 1-19.
- Ryan, D. M., Bonnett, D. M., & Gass, C. B. (2006). Sobering thoughts: Town hall meetings on fetal alcohol spectrum disorders. American Journal of Public Health, 96(12), 2098-2101.
- Ryan, S., & Ferguson, D. L. (2006). On, yet under, the radar: students with fetal alcohol spectrum disorder. Exceptional Children, 72(3), 363-379.
- Wingood, G. M., & DiClemente, R. J. (2008). The ADAPT-ITT model: a novel method of adapting evidence-based HIV Interventions. JAIDS Journal of Acquired Immune Deficiency Syndromes, 47, S40-S46.